CLINICAL TRIAL: NCT01165086
Title: Reducing Dietary Energy Density by Incorporating Vegetables in Order to Decrease Energy Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Principle Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: FoodED101; R37DK039177 (NIH); R01DK059853 (NIH)
Record Dates: First submitted 2010-07-16; First posted 2010-07-19 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Other: Incorporating vegetables into the diet to reduce energy density — The entree portion of breakfast, lunch, and dinner meals will be manipulated to be a standard energy density, a 15% reduction in energy density, or a 25% reduction in energy density.

SUMMARY:
This study will test the hypothesis that incorporating vegetables into meals as a method of reducing the energy density will result in increased vegetable intake and decreased energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20-45 years

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Energy intake | 3 weeks

SECONDARY OUTCOMES:
Vegetable intake | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Blatt AD, Roe LS, Rolls BJ. Hidden vegetables: an effective strategy to reduce energy intake and increase vegetable intake in adults. Am J Clin Nutr. 2011 Apr;93(4):756-63. doi: 10.3945/ajcn.110.009332. Epub 2011 Feb 2. PMID 21289225